CLINICAL TRIAL: NCT04015791
Title: Clinical Evaluation of NOCISCAN-Lumbar Spine (LS) Disc MR Spectroscopy (MRS) for Diagnosis of Discogenic Low Back Pain and Correlation With Surgical Outcomes
Brief Title: NOCISCAN-Lumbar Spine (LS) Clinical Evaluation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nocimed, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: NM005
Record Dates: First submitted 2019-06-29; First posted 2019-07-11 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Disc Disease
Keywords: lumbar disc disease; MR Spectroscopy; Nociscan
MeSH Terms: conditions — Intervertebral disc disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Match Group: Surgery conducted at the disc level corresponding with the highest level of NOCISCORE value in the subject and that is classified as either NOCI + or NOCI mild
  Interventions: Other: NOCISCAN-LS Disc MR Spectroscopy
- Miss Group: Surgery conducted at a disc that: (a) corresponds with a low relative NOCISCORE value in the subject and that is classifies as NOCI - or (b) excludes the disc level with the highest NOCISCORE value in the subject and that is classifies as NOCI+ or NOCI mild
  Interventions: Other: NOCISCAN-LS Disc MR Spectroscopy

INTERVENTIONS:
Other: NOCISCAN-LS Disc MR Spectroscopy — The investigational Nociscan Suite is a software suite that works with existing high field MR systems and MRS pulse sequence via and optimized protocol to conduct MRS exam of lumbar discs. The software suite post-processes the NOCISCAN-LS disc MRS exam data to calculate ratios of spectroscopic signals at regions along the MRS frequency spectrum associated with certain chemicals that change with degeneration and pain
  Other Names: MR Spectroscopy (MRS)

SUMMARY:
A prospective, double blinded, multi-center study to assess the validity and clinical utility of the pre-operative NOCISCAN-LS software in the identification of painful lumbar discs, and the correlation with improved surgical outcomes at 3, 6, 12 and 24 months (follow-up) following spine surgery in a single enrollment arm of subjects with chronic symptomatic single level degenerative disc disease (DDD) at L3 to S1, but with two evaluation groups- Match Group and Miss Group,of subjects based on the association between the NOCISCORE results of treated and untreated disc levels.

ELIGIBILITY:
Inclusion Criteria:

1. Has history consistent with degenerative disc disease as noted by back pain of discogenic origin with or without leg pain
2. Has one of more of the following conditions as documented by CT or MRI and plain X-rays:

   1. Modic changes
   2. High intensity zones in the annulus
   3. Loss of discogenic height
   4. Decreased hydration of the disc
3. Has single level symptomatic degenerative involvement from L3 to S1 in which surgical treatment is indicated
4. Skeletally mature male or female (non-pregnant) between 18 and 70 years of age
5. Pre-operative score ≥ 40% on Oswestry Disability Index
6. VAS back pain score ≥ 40 mm and that is greater than the VAS leg pain scores
7. Patient has failed at least ≥6 months of non-operative treatment that may have included physical therapy, bed rest, anti-inflammatory or analgesic medications, chiropractic care, acupuncture, massage therapy or home-directed lumbar exercise programs
8. In subject who receives pre-operative provocative discography (PD), the PD was performed more than 6 week prior to the scheduled NOCISCAN- LS Exam OR Is scheduled to be conducted after the Nociscan exam
9. Subject is willing to sign an Institutional Review Board approved Informed Consent and HIPAA Authorization forms, and is physically and mentally able to complete study forms and otherwise willingly adhere to the requirements of the protocol in the opinion of the investigator

Exclusion Criteria:

1. Has primary diagnosis of spinal condition other than degenerative disc disease at the involved level;
2. Has had prior lumbar back surgery or intradiscal treatments at any lumbar level (Note: diagnostic provocative or anesthetic discography are not excluded; micro-discectomy +- laminectomy patients greater than 6 months postop are not excluded)
3. Surgery planned at more than one level
4. Radiographic evidence of clinically relevant lumbar vertebral abnormalities, including

   * Greater than Grade 1 spondylolisthesis according to Meyerding classification at the involved level;
   * Any posterior lumbar element insufficiency (e.g. Spondylolysis, pars fracture, or prior facet resection;
   * Lumbar scoliosis with a Cobb angle of greater than 11 degree
   * Symptomatic kyphosis or flat black syndrome
   * Evidence of prior fracture or trauma to the L1, L2,L3, L4 or L5 levels in either compression or burst; Note: Modic end plate changes will not be excluded
5. Radiographic evidence of lumbar disc herniation with extrusion
6. Clinically significant spinal canal stenosis as assessed by the Investigator
7. Any significant motor strength deficit in lower extremities
8. Suspicion of Sacro Iliac and/ or Facet joint pain as the primary pain generator;
9. Has a condition that requires post-operative medications that interfere with fusion, such as immunosuppressive drugs, steroids or prolonged use of non-steroidal anti-inflammatory drugs. This does not include low dose aspirin for prophylactic anticoagulation
10. Has active bacterial infection, either local or systemic and/or potential for bacteremia
11. Has presence of active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin) during the past 5 years
12. Chronic disease (other than degenerative disc disease), chronic pain syndrome (other than discogenic low back pain), or psychological dysfunction, which may , in the opinion of the Investigator compromise a subject's ability to comply with study procedures, and/ or may confound data;
13. Applicable exclusionary criteria for standard lumbar MRI exam;
14. Has pending litigation, except where required by the insurer as condition of coverage;
15. BMI > 40kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 240 subjects that are approved and scheduled for surgery at a single level from L3 to S1 to treat chronic, severe, primary axial, discogenic, low back pain via maximum of 14 sites
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index Assessment to assess improvement in lumbar pain | 24 months
  Oswestry Disability Index is an index derived from Oswestry Low Back Pain Questionnaire used in several studies to quantify disability for low back pain. Each of the 10 items is scored from 0-5. The maximum score is therefore 50. This will be completed at 12 month follow up to see if there is an improvement of at least 15 points at 12 months Follow-up for Match Group versus Miss Group subjects. Mean Oswestry Disability Index score changes at 3, 6 and 24 months post-operative follow-up will be evaluated for Match versus Miss Group

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) to assess the intensity of pain | 2 years
  Visual Analog Scale for pain is a validated tool used in determining the subjective level of pain in an individual. It will be completed at Mean Visual Analog Scale score changes for back pain at 3,6, 12 and 24 months post-op follow up for Match versus Miss Group
Demonstrate correlation of NOSCISCORE results to Provocative Discography +/- results in subset of study subjects that receive pre-operative provocative discogram | 24 months
  Compare NOCISCORE results for Provocative discography positive discs versus Provocative discography negative discs in study subjects receiving pre-operative discogram

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Back Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided